CLINICAL TRIAL: NCT03819309
Title: Efficacy of Transvaginal Ultrasound-guided Aspiration for Treatment of Tubo-ovarian Abscess Compared With Laparoscopy
Acronym: PACTOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K170917J
Record Dates: First submitted 2019-01-17; First posted 2019-01-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Uncomplicated Tubo Ovarian Abscess
Keywords: tubo ovarian abscess; transvaginal aspiration; laparoscopy
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided transvaginal drainage (Experimental): evacuation of the TOA will be done by ultrasound-guided transvaginal puncture under simple sedation or under general anesthesia if necessary
  Interventions: Procedure: Ultrasound-guided transvaginal drainage
- Laparoscopy (Active Comparator): TOA will be evacuated by coelioscopy under general anesthesia
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Ultrasound-guided transvaginal drainage — evacuation of the TOA will be done by ultrasound-guided transvaginal puncture under simple sedation or under general anesthesia if necessary
  Arms: Ultrasound-guided transvaginal drainage
Procedure: Laparoscopy — TOA will be evacuated by coelioscopy under general anesthesia
  Arms: Laparoscopy

SUMMARY:
"Tubo-ovarian abscess (TOA) include pyosalpinx, ovarian abscess, tubo-ovarian abscess and Douglas abscess. The only randomized study evaluating TOA treatment reported a higher cure rate (90 versus 65%) when antibiotic therapy is associated with abscess evacuation.

TOA evacuation can be performed by surgery or by drainage. No studies have compared success rates between those two methods.

Concerning surgery, current practices recommend performing laparoscopy which allows a shorter hospital stay, a lower complication rate and high success rates.

The majority of published studies reporting radiological drainage concern ultrasound-guided transvaginal drainage. The reported success rates range from 77 to 100%. The PACTOL trial is a randomized, prospective, controlled, open, parallel, non-inferiority, multicenter trial comparing the efficacy of transvaginal drainage versus laparoscopy in both arms with antibiotic therapy in the treatment of TOA.

DETAILED DESCRIPTION:
"Tubo-ovarian abscess (TOA) include pyosalpinx, ovarian abscess, tubo-ovarian abscess and Douglas abscess from genital organs.

The only randomized study evaluating TOA treatment reported a higher cure rate (90 versus 65%) when antibiotic therapy is associated with abscess evacuation.

This TOA evacuation can be performed by surgery or by drainage. No studies have compared, even retrospectively, success rates between those two methods.

Current practices recommend performing conservative surgery by laparoscopy which allows a shorter hospital stay, a lower complication rate and high success rates (90%).

The majority of published studies reporting radiological drainage concern ultrasound-guided transvaginal drainage. The reported success rates range from 77 to 100%.

Thus, the literature supports the association antibiotic / evacuation of the TOA (surgical or drainage) because of a high success rate. However, there is no comparative data to favor laparoscopic evacuation over transvaginal drainage.

The French recommendations for the management of TOA recommend the use of transvaginal drainage or laparoscopy for the treatment of ATO always in combination with antibiotics. The recommended antibiotic treatment combines triantibiotherapy with doxycycline, cephalosporin and metronidazole.

The main objective of the PACTOL trial will be to demonstrate non-inferiority of the transvaginal approach in the treatment of ATO versus laparoscopy in terms of efficacy. The secondary objective of our study is to confirm the less invasive nature of transvaginal drainage (reduction of hospital stay, reduction of hospital costs and better tolerance).

The PACTOL trial is a randomized, prospective, controlled, open, parallel, non-inferiority, multicenter trial comparing the efficacy of transvaginal drainage versus laparoscopy in both arms with antibiotic therapy in the treatment of TOA.

Interventions The PACTOL trial will compare two techniques of TOA evacuation : transvaginal drainage and laparoscopy drainage. In both cases, preoperative anesthesic consultation will be performed. All included patients will be hospitalized and treated with intravenous antibiotics according of French national guidelines. The TOA evacuation will be performed according to the result of randomization within 3 days of hospitalization.

Each patient will be included after receiving consent to participate in the study. After inclusion, randomization will be performed with two parallel arms:

* arm A : intravenous probabilistic triantibiotherapy + TOA drainage by transvaginal drainage under ultrasound control.
* Arm B : intravenous probabilistic triantibiotherapy + TOA drainage by laparoscopy.

The computerized randomization procedure will be performed before the surgery. The randomization should take place maximum 3 days after the beginning of the antibiotic treatment.

In both arms, a probabilistic triantibiotherapy known as a reference for the treatment of TOA in genital infection will be delivered as soon as the patient is hospitalized.

This triantibiotherapy will be composed by Ceftriaxone 1 to 2g x1 per day + Metronidazole 500 mg x3 per day + Doxycycline 100 mg x2 per day intravenously initially then per os and intramuscular for 21 days.

In case of allergy, alternatives may be Ofloxacin 400 mg x 2 per day + Metronidazole 500 mg x 3 per day IV for 21 days or Cefoxitin 1 to 2 gx 3 per day + Doxycycline 100 mg x 2 per day IV for 21 days according to the recommendations of the CNGOF.

Arm A : Transvaginal drainage:

The patient will be managed in the operating room, with simple sedation, in lithotomy position. If the patient is not comfortable, a general anesthesia will be performed.

The operator (a senior physician) will use pelvic ultrasound by the endovaginal route to identify TOA. The content of the abscess will be aspirated using a syringe and will be sent for bacteriological analysis.

Arm B : Laparoscopy:

The patient will be managed in the operating room, under general anesthesia. The surgical approach will be laparoscopic. The operator (a senior doctor) will report the inventory of the pelvis and abdomen. The TOA will then be located and evacuated with a collection of the drainage liquid to send it for bacteriological analysis.

Conservative treatment will be recommended but left to the discretion of the operator. After complete drainage and washing of the pelvic cavity, the procedure will be completed. Drainage by redon left in place will be recommended but also left to the choice of the operator.

Examination on inclusion The initial assessment will be performed in the hospital emergency by a gynecologist. Patient's hemodynamic variables (heart rate, blood pressure, temperature) will be recorded and signs of shock sought. The pelvic examination will include an abdominal palpation, speculum examination searching for leucorrhoea, metrorrhagia, cervical examination, vaginal and endocervical sampling for chlamydia, gonococci, mycoplasma. Vaginal examination looking for pain during uterine mobilization, lateralized pain in the vaginal sac and lateral uterine mass will be performed.

Biological tests searching for inflammatory syndrome, urinary infection, pregnancy test as well as preoperative tests will be performed.

Pelvic ultrasound for the diagnosis of TOA will be performed using suprapubic and endovaginal routes with 2 baseline measurements in the sagittal plane and a measurement in the axial plane of the latero-uterine mass. If there is doubt about the diagnosis, performing a CT or MRI is allowed.

The inclusion and non-inclusion criteria will be verified by gynecologist. Details of the protocol will be provided to the patient through a written notice and oral explanations. Signed consent forms will be collected from patients agreeing to participate in the study prior to enrollment, by a senior gynecologist acting as a local investigator in the trial. The patient will be informed of the possibility of using her data for a future fertility study.

Each patient will be included after receiving consent to participate in the study.

Randomization Once the patient has been informed, informed consent obtained and the criteria for inclusion and exclusion have been checked, a single-blind randomization with a 1:1 ratio will be performed electronically with a secure internet platform (CleanWeb) .

The randomization list will be generated by computer, stratified per center, with blocks of different sizes. The day of the randomization will be considered as the beginning of follow-up (D0).

Patients will be randomized during their hospitalization, during the inclusion visit.

Given the nature of the intervention, health professionals and patients cannot be blinded to the randomization group. However, the evaluation of the primary endpoint will be done by the statistician who will be blind to the treatment received by each patient.

Intrahospital management During their stay in hospital, the patients will be managed according to the standard practice of the center.

In hospital, according to the usage, a monitoring of the temperature, the arterial pressure, the heart rate, the saturation will be carried out every 6 hours.

A clinical examination by a gynecologist will be carried out daily to follow up the infection and to detect possible complications secondary to treatment. During this evaluation, the pain will be quantified using a visual analogue scale the next day and 3 days after the TOA evacuation. The EQ-5D questionnaire and a standardized surgical report will also be given to the patient during this consultation.

Postoperative consultation For the determination of the primary outcome, an ultrasound and postoperative consultation are planned at 6 weeks of hospitalization +/- 2 weeks. This consultation will

* inform if a reintervention (transvaginal drainage, laparoscopy or laparotomy) or a new antibiotic treatment were necessary to treat a recurrence of TOA since discharge from hospital. The practitioner will look for a recurrence of TOA through the clinical examination.
* report any post-operative complications that will be classified according to the Clavien-Dindo classification.
* inform the patient's desire and plan to obtain a pregnancy during the next two years in order to decide to include the patient in the evaluation of fertility after treatment of an TOA by comparing transvaginal drainage and laparoscopy. Patients with a pregnancy desire will be informed that TOA can be complicated by infertility. Then, patients with difficulties in procreation can be offered a diagnostic laparoscopy to find a cause of infertility, depending on the etiological assessment.

Follow up Patients who will not attend the postoperative consultation will be contacted by phone to collect data regarding possible recurrence of TOA and postoperative complications. If the patient does not attend a scheduled appointment, she will be contacted by phone to arrange a new appointment. For this, a record of his personal details (name, phone, availability) will be kept in her medical file. After 3 phone call attempts (different days and time slots), the patient will be considered lost to follow-up.

After their initial postoperative consultation, patients will attend follow up 2 years for those who had a pregnancy desire. These one will be contacted by phone 24 months after their beginning of follow-up.

Patients will have follow-up in the form of a phone interview or self-administered questionnaire sent by email or mail (depending on patients preference) 2 years after drainage of the abscess to assess the secondary criterion of pregnancy rate."

ELIGIBILITY:
"Inclusion criteria :

* Major patient aged ≤ 50 at the time of inclusion
* Patient hospitalized for TOA diagnosis defined by:

  * a high genital infection (major criteria of recommendations for the clinical practice of CNGOF): spontaneous pelvic pain and induced adnexal pain and / or uterine mobilization pain;
  * Visible ultrasound collection in the form of a latero-uterine mass measuring at least 3 cm detailed in the recommendations of the CNGOF:

    * tubal wall thickening> 5 mm
    * OR sign of the gear wheel (thickened tubal fringes giving an incomplete septa appearance)
    * OR Heterogeneous lateral mass + / - compartmentalized with fine echoes
* Biological inflammatory syndrome (defined by CRP> 20 or white blood cell> 10,000 / mm3)
* Uncomplicated: good hemodynamic tolerance, not broken

Exclusion criteria :

* Suspected malignant tumor or Borderline
* Complicated abscess: abscess rupture, generalized peritonitis, septic shock
* Known HIV infection with CD4 count <200 / mm3, immunosuppression
* Patient already operated for TOA in progress
* TOA not accessible to vaginal puncture
* Multiple antecedents of abdominal surgeries that make it more difficult to surgically access the abdominopelvic cavity
* Pregnancy in progress or breastfeeding
* Patient with a contraindication to general anesthesia
* Poor understanding of the French language
* Patient under guardianship or curatorship
* Patient under AVK without relay by LMWH possible
* Known allergies or contraindications to any of the drugs used in the research
* Patient participating in another interventional research protocol
* No affiliation to the social security scheme or the CMU (universal health cover)
* Absence of informed consent, written and signed"

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Cure rate | 6 weeks
  "The cure rate is defined by a composite criterion at 6 weeks of the procedure:
  * No reoperation (puncture or coelioscopy) for TOA
  * No reintroduction of antibiotic therapy for TOA
  * Absence of latero uterine collection ≥ 3 cm on ultrasound"

SECONDARY OUTCOMES:
Number of days of hospital stay | 6 weeks
Costs related to the hospital care of ATO at 6 weeks | 6 weeks
Pregnancy rate in patients under 45 years of age at 2 years | 2 years
Number of intra uterine pregnancy | 2 years
Number of extra uterine pregnancy | 2 years
Number of term of delivery | 2 years
Number of spontaneous pregnancy | 2 years
Number of pregnancy after tubal surgery | 2 years
Number of pregnancies obtained by in vitro fertilization | 2 years
Health-related quality of life self-report mesured by EuroQol 5 Dimention | at baseline and at 6 weeks
Rate of per operative complications (at 6 weeks) grade ≥ 2 (Clavien-Dindo classification) | 6 weeks
Rate of postoperative complications (at 6 weeks) grade ≥ 2 (Clavien-Dindo classification) | 6 weeks
Pain self-assessment mesured by Visual Analog Scale the next day and 3 days after evacuation | the next day and 3 days after evacuation
numbers of adverse events | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin Koskas, M.D. Ph.D., Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided